CLINICAL TRIAL: NCT00970138
Title: A Randomized Phase 2/3 Study of Apatinib as Third Line Treatment in Patients With Metastatic Gastric Carcinoma
Brief Title: Apatinib Versus Placebo as a Third Line Treatment in Patients With Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Jin Li/Dr, Fudan University cancer hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009APA-MGC
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2010-09

CONDITIONS: Gastric Carcinoma
Keywords: Progress free survival; Toxicity; Response rate; Overall survival; Quality of live
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A 850 (Experimental): apatinib 850 mg qd, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: apatinib tablet
- B 425 (Experimental): apatinib 425 mg bid, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: apatinib tablet
- C pla (Placebo Comparator): placebo bid, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: apatinib tablet

INTERVENTIONS:
Drug: apatinib tablet — A850: apatinib 850 mg qd p.o. plus placebo qd p.o. until disease progression or intolerable toxicity or patients withdrawal of consent
  B425: apatinib 425 mg bid p.o. until disease progression or intolerable toxicity or patients withdrawal of consent
  Cpla: placebo bid p.o. until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
Apatinib is a tyrosin-inhibitor agent targeting at vascular endothelial growth factor receptor (VEGFR), and it's anti-angiogenesis effect has been viewed in preclinical tests. The investigators' phase I study has shown that the drug's toxicity is manageable and the maximum tolerable daily dose is 850 mg. The purpose of this study is to determine whether apatinib can improve progression free survival compared with placebo in patients with metastatic gastric carcinoma who failed two lines of chemotherapy.

DETAILED DESCRIPTION:
Up to now, although FU based, cisplatin based and taxane based regimen, and ECF regimen have been suggested as the first line therapy for A/MGC by FDA, the efficacy of these treatment is still unsatisfied for their toxicity and limitation in prolonging survival. Based on the promising results of apatinib in the phase I study, this clinical trial has been designed to evaluate whether apatinib can improve progression free survival in patients with metastatic gastric carcinoma who failed two lines of chemotherapy compared with placebo. Patients will be randomized to 3 groups, one group patients will receive the treatment of apatinib 850mg qd, one group patients will receive apatinib 425mg bid, and the other group will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 70 years of age
* Histologically confirmed advanced or metastatic adenocarcinoma of the stomach
* Have failed for 2 lines of chemotherapy
* Life expectancy of more than 3 months
* ECOG performance scale ≤ 2
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin
* More than 4 weeks for operation or radiotherapy
* More than 4 weeks for cytotoxic agents or growth inhibitors
* Adequate hepatic, renal, heart, and hematologic functions (platelets > 80 × 109/L, neutrophil > 2.0 × 109/L, serum creatinine ≤ 1.5mg/dl, total bilirubin within upper limit of normal(ULN), and serum transaminase≤2.5×the ULN).

Exclusion Criteria:

* Pregnant or lactating women
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Any factors that influence the usage of oral administration; Evidence of CNS metastasis
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Intercurrence with one of the following: hypertension, coronary artery disease, arrhythmia and heart failure
* Receiving the therapy of thrombolysis or anticoagulation
* Abuse of alcohol or drugs
* Allergy to the ingredient of the agent or more than two kinds of food and drug
* Less than 4 weeks from the last clinical trial
* Disability of serious uncontrolled intercurrence infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 8 weeks

SECONDARY OUTCOMES:
Overall survival safety | 8 weeks
DCR (Disease control rate) | 8 weeks
ORR (Objective response rate) | 8 weeks
QoL (Quality of life) | 8 weeks
Toxicity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952